CLINICAL TRIAL: NCT02877121
Title: Respiratory Muscle Function and Neural Respiratory Drive in Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Zhang Jianheng (Other)
Responsible Party: Sponsor-Investigator, Zhang Jianheng, Dr, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: gird2016
Record Dates: First submitted 2016-08-10; First posted 2016-08-24 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-08

CONDITIONS: State Key Laboratory of Respiratory Disease
Keywords: interstitial lung disease; Respiratory Muscle Function; Neural Respiratory Drive
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the Respiratory Muscle Function and Neural Respiratory Drive in Interstitial Lung Disease patients.

DETAILED DESCRIPTION:
In total, 50 patients with interstitial lung disease (ILD) are going to recruited.The patients are studied at the afternoon in a semirecumbent position. After the application of topical anaesthesia (2% xylocaine), the patient will be asked to swallow two balloon-tipped catheters and the multi-pair esophageal electrode catheter through the nose into the their right position.

At the first period, the stable signals of unassisted spontaneous breathing (about 10min) were chosen to be recorded. The Esophageal and gastric balloon-catheters are used to detect the intra-thoracic and abdominal pressure.The diaphragm electromyogram (EMGdi) will be recorded from a multipair esophageal electrode.The baseline data of the respiratory muscle activity will be detected by these catheters and electrode.p0.1 (the negative airway pressure generated during the first 100 ms of an occluded inspiration) will be also meassured.

After the first period, the nonvolitional tests on respiratory muscle function and strength (twitch mouth and transdiaphragmatic pressure during bilateral magnetic phrenic nerve stimulation (TwPmo and TwPdi) will be done.

After the second period,the patients will be ask to perform different maneuvers, including maximal inspiration against a closed valve ,maximal inspiration to total lung capacity (TLC),maximalexpiration at the total lung capacity (TLC) against a closed valve and maximal sniff from functional residual capacity(FRC).Each maneuver will repeated more than three times with an interval of 30 s or more. Inspiratory capacity(IC),global maximal inspiratory pressure (PImax), maximal sniff nasal pressure (SnPna) and maximalexpiratory pressure will be meassured with the balloon-catheters.The maximal value of the diaphragm electromyogram (EMGdi) will be recorded during these maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial lung disease patient meet the diagnose criteria of interstitial lung disease

Exclusion Criteria:

1. Severe Cardiovascular disease
2. Pneumonia
3. Neuromuscular and chest wall deformity
4. Respiratory arrest
5. Cardiovascular instability (hypotension, arrhythmias, myocardial infarction)
6. Change in mental status; uncooperative patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial Lung Disease patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
transdiaphragmatic pressure during bilateral magnetic phrenic nerve stimulation (5-20cmH2O)(TwPdi) | 20-30minutes

SECONDARY OUTCOMES:
the The diaphragm electromyogram (EMGdi)(10-300uv ) | 20-30minutes
the negative airway pressure generated during the first 100 ms of an occluded (p0.1)(from -0.5 to -5cmH2O) | 20-30minutes
The global maximal inspiratory pressure (PImax) of the Interstitial Lung Disease | 20-30minutes
The maximal sniff nasal pressure (SnPna)of the Interstitial Lung Disease patients(5-100cmH2O) | 20-30minutes
The maximalexpiratory pressure (MEP)of the Interstitial Lung Disease patients(5-100cmH2O) | 20-30minutes
The twitch mouth and during bilateral magnetic phrenic nerve stimulation (TwPmo)(from -2 to-20cmH2O) | 20-30minutes

CONTACTS AND LOCATIONS:
Locations (1):
- TheFirst Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided